CLINICAL TRIAL: NCT04700748
Title: Diffusion-weighted MRI to Predict Treatment Response in Stereotactic Radiotherapy of CNS Metastases
Brief Title: Diffusion-weighted MRI to Predict Treatment Response in Stereotactic Radiotherapy of Central Nervous System (CNS) Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MR-SRS-001
Record Dates: First submitted 2020-12-28; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Radiotherapy; Brain Metastases; Sensitivity; Radionecrosis
Keywords: Diffusional variance decomposition; DIVIDE; Brain metastasis; Radiation treatment; Treatment response; Radionecrosis; Radiation damage; Radiation sensitivity; Magnetic resonance imaging
MeSH Terms: conditions — Brain Neoplasms; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diffusion-weighted MRI to predict treatment response in stereotactic radiotherapy of CNS metastases. (Other): Patients with brain metastases who will receive radiotherapy to the brain will undergo diffusion-weighted magnetic resonance imaging (MRI) at the same time as dose planning MRI is performed, after end of radiotherapy, and after 3 and 6 months after end of radiotherapy.
  Interventions: Radiation: Brain metastases radiation

INTERVENTIONS:
Radiation: Brain metastases radiation — Brain metastases radiation according to clinical practice.

SUMMARY:
Stereotactic radiation therapy is an important and common method of treating brain metastases in patients with malignant disease. Today, however, there are no methods available to determine the metastasis' radiation sensitivity in advance and treatment responses can only be seen by changing of the size of the metastasis on conventional X-ray examinations, computed tomography (CT) and magnetic resonance imaging (MRI). Changes in the size of the metastases is something that is often seen weeks / months after treatment is completed. At Lund University Hospital, a new imaging technique, diffusional variance decomposition (DIVIDE), has now been developed. With this technique, the scatter in isotropic and anisotropic diffusion can be measured for each measuring point, which provides significantly more information about the properties of the tissue compared to current methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients prescribed stereotactic radiation therapy to the brain, where MRI imaging is included in the treatment preparations.
2. Cohesive remaining solid tumor component of ≥10mm.
3. Age ≥18 years.
4. World Health Organisation (WHO) performance status 0-1.

Exclusion Criteria:

1. Inability to decide for oneself on participation in the study.
2. Inability to understand the Swedish language.
3. Metastases close to the base of the skull.
4. Contraindications to conducting an MRI examination.
5. Contraindications to obtaining contrast media during MRI examination.
6. Expected survival less than 6 months.
7. Previous radiation treatment to the same site in the brain, i.e. current treatment is a rope radiation.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Grade of radiation sensitivity to brain metastasis. | Is evaluated after end of radiotherapy, that is after 3 days, as all subjects receive 3x10 Gy.
  Evaluation done by MRI to see whether radiation sensitivity can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Grade of radiation sensitivity to brain metastasis. | Is evaluated after 3 months after end of treatment.
  Evaluation done by MRI to see whether radiation sensitivity can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Grade of radiation sensitivity to brain metastasis. | Is evaluated after 6 months after end of treatment.
  Evaluation done by MRI to see whether radiation sensitivity can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Early changes in the tumor during and after completion of radiation therapy. | Is evaluated after end of radiotherapy, that is after 3 days, as all subjects receive 3x10 Gy.
  Evaluation done by MRI to see whether early changes in the tumor can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Early changes in the tumor during and after completion of radiation therapy. | Is evaluated after 3 months after end of treatment.
  Evaluation done by MRI to see whether early changes in the tumor can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Early changes in the tumor during and after completion of radiation therapy. | Is evaluated after 6 months after end of treatment.
  Evaluation done by MRI to see whether early changes in the tumor can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Changes linked to treatment responses. | Is evaluated after end of radiotherapy, that is after 3 days, as all subjects receive 3x10 Gy.
  Evaluation done by MRI to see whether changes in the tumor can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Changes linked to treatment responses. | Is evaluated after 3 months after end of treatment.
  Evaluation done by MRI to see whether changes in the tumor can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Changes linked to treatment responses. | Is evaluated after 6 months after end of treatment.
  Evaluation done by MRI to see whether changes in the tumor can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Differentiate between radiation damage (radionecrosis) and residual / recurrent tumor. | Is evaluated after end of radiotherapy, that is after 3 days, as all subjects receive 3x10 Gy.
  Evaluation done by MRI to see whether differentiation between radionecrosis and residual/recurrent tumor can be measured during radiotherapy and after 3 and 6 months after end of treatment.
Differentiate between radiation damage (radionecrosis) and residual / recurrent tumor. | Is evaluated after 3 months after end of treatment.
  Evaluation done by MRI to see whether differentiation between radionecrosis and residual/recurrent tumor can be measured during radiotherapy after 3 months after end of treatment.
Differentiate between radiation damage (radionecrosis) and residual / recurrent tumor. | Is evaluated after 6 months after end of treatment.
  Evaluation done by MRI to see whether differentiation between radionecrosis and residual/recurrent tumor can be measured during radiotherapy and after and 6 months after end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No